CLINICAL TRIAL: NCT06601205
Title: A Randomized, Phase IIB, Double Blind, Placebo Controlled, Multicenter, Pre-surgical, Window-of-opportunity Trial of Finasteride Vs. Low-dose Flutamide Vs. Placebo in Prostate Cancer (2F Trial)
Brief Title: Finasteride and Flutamide in Pre-surgical Trial in Prostate Cancer.
Acronym: 2F
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Universita degli Studi di Genova (Other); Cliniche Humanitas Gavazzeni (Other); Università Politecnica delle Marche (Other); European Institute of Oncology (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Director of Medical Oncology Division, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13CE20102003; Italian League against Cancer (Other: LILT (Lega Italiana contro i Tumori)); Berlucchi Foundation (Other: Fondazione Berlucchi)
Record Dates: First submitted 2019-02-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer; Prostatic Intraepithelial Neoplasia
Keywords: Prostate Cancer; Prostatic Intraepithelial Neoplasia; Chemoprevention; Flutamide; Finasteride; Biomarkers, drug response; Karyometry
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Intraepithelial Neoplasia | interventions — Flutamide; Finasteride

STUDY DESIGN:
Intervention Model Description: The study was a prospective, randomized, phase IIB, placebo controlled, double-blind, pre-surgical trial of Finasteride 5 mg day versus Flutamide 250 mg day versus placebo in men with PCa. Patients with a biopsy proven, clinically intracapsular prostate cancer who were candidate to radical retropubic prostatectomy were enrolled in four different institutions in Northern Italy. Different biopsy criteria according to each contributing centre were acceptable provided that a minimum of 8 cores were evaluable. Patients were randomized to receive either flutamide, 250 mg/day orally, or finasteride, 5 mg/day orally, or oral placebo in a double-blind manner beginning 4 to 6 weeks before surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drugs and placebo were purchased through the Galliera Hospital Pharmacy, encapsulated to preserve blinding, then packaged and labelled for the study under GMP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Flutamide (Experimental): 1 tablet 250 mg daily until the day before surgery
  Interventions: Drug: Flutamide
- Finasteride (Experimental): 1 tablet 5 mg daily until the day before surgery
  Interventions: Drug: Finasteride
- Placebo (Placebo Comparator): 1 tablet daily until the day before surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Flutamide — 1 tablet daily until the day before surgery
  Other Names: Arm A
  Arms: Flutamide
Drug: Finasteride — 1 tablet daily until the day before surgery
  Other Names: Arm B
  Arms: Finasteride
Other: Placebo — 1 tablet daily until the day before surgery
  Other Names: Arm C
  Arms: Placebo

SUMMARY:
Pre-surgical, window-of-opportunity trials provide a suitable model to assess the activity of preventive interventions in a cost-effective manner using tissue biomarkers as surrogate endpoints. Finasteride has been shown to reduce prostate cancer development in a large phase III trial, and flutamide has a well-known anticancer effect in advanced prostate cancer at the dose of 750 mg/day.

DETAILED DESCRIPTION:
In this randomized, phase IIB, double blind, placebo controlled, multicenter, pre-surgical, window-of-opportunity trial we compared the effects of finasteride (5 mg/day) versus low-dose flutamide (250 mg/day) or placebo on tissue biomarkers in patients with prostate cancer who were candidate to radical surgery. Specifically, the effects of both drugs on the change in epithelial cell nuclear area in prostate cancer tissue between pre- and post-treatment biopsies was evaluated (primary endpoint). Moreover, the changes of the proliferation marker Ki-67 and of karyometric parameters in benign, dysplastic (HG-PIN) and malignant tissues were evaluated (secondary endpoints). Additional endpoints include the changes of serum PSA and testosterone, assessment of toxicity, overall survival, recurrence-free survival and event-free (recurrence + death) survival. Patients with intracapsular biopsy proven prostate cancer were randomized to either flutamide, 250 mg/day, or finasteride, 5 mg/day, or placebo for 4-6 weeks before radical prostatectomy. Blood samples were taken before and after treatment. At surgery, end-of-study ex-vivo biopsies were obtained from the prostatectomy specimens to assess the treatment changes in nuclear area (primary endpoint), Ki-67, topoisomerase-II-α and a 20-feature karyometric discrimant function in normal, high-grade PIN and malignant tissue. After surgery patients were followed up for at least 15 years to assess recurrence and/or mortality. We also plan to follow-up patients by telephone interview to assess their vital status for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Patients with a biopsy proven, clinically intracapsular PCa who are candidates to radical retropubic prostatectomy
* ECOG performance status ≤ 2
* Satisfactory hematological and biochemical functions:

  * Platelets ≥100 x 10^9/L
  * AST and ALT in the normal range
* Able to understand and sign an informed consent

Exclusion Criteria:

* Previous hormone treatment during the 8 weeks before enrollment
* Neurologic and psychiatric diseases precluding patient participation in the study
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing or participating in the study and/or comply with the study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2008-03-20 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Change of Nuclear area size | 4-6 weeks (baseline and at the end of the study biopsy)
  The study primary endpoint is the change of epithelial cell nuclear area in prostate cancer tissue and HG-PIN tissue between pre- and post-treatment measure in the two active treatment arms (Finasteride or Flutamide) compared with the placebo arm.

SECONDARY OUTCOMES:
Change of ki-67 value | 4-6 weeks (baseline and at the end of the study biopsy)
  Changes of Ki-67 labeling index in normal, HG-PIN and prostate cancer cells in the three arms.
Change Kariometry value | 4-6 weeks (baseline and at the end of the study biopsy)
  Changes in karyometric features in normal HG-PIN and prostate cancer cells in the three arms.
Serum biomarkers values | 4-6 weeks (on blood samples at baseline and the day before surgery)
  Changes in total PSA, free PSA and testosterone concentrations after treatment in the three arms.
Adverse Events | 4-6 weeks (during the treatment)
  Toxicity is assessed using the National Cancer Institute-Common Terminology Criteria for Adverse Events (version 3, 2003).
Recurrence-free survival | up to 20 years
  Comparison of Recurrence-free survival among arms will be assessed by the Kaplan Meier actuarial survival curves and analyzed by the log-rank test and the Cox proportional hazard model for multivariate analyses. Vital status and medical condition will be assessed by telephone interview and clinical visit.
Comparison of Event free survival | up to 20 years
  Comparison of Event free survival among arms will be assessed by the Kaplan Meier actuarial survival curves and analyzed by the log-rank test and the Cox proportional hazard model for multivariate analyses. Vital status and medical condition will be assessed by telephone interview and clinical visit.
Comparison of Overall Survival | up to 20 years
  Comparison of Overall Survival among arms will be assessed by the Kaplan Meier actuarial survival curves and analyzed by the log-rank test and the Cox proportional hazard model for multivariate analyses. Vital status and medical condition will be assessed by telephone interview and clinical visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, MD, Principal Investigator — E.O. Ospedali Galliera
Locations (1):
- Medical Oncology Ente Ospedaliero Ospedali Galliera, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: No